CLINICAL TRIAL: NCT06486454
Title: Real-world Evaluation of the HistoSonics Edison System for Treatment of Liver Tumors Across Multidisciplinary Users (BOOMBOX: Master Study)
Status: Recruiting | Type: Observational
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP3828
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Liver Neoplasms; Primary Liver Cancer; Secondary Liver Cancer; Tumor Liver; Benign Liver Tumor
Keywords: histotripsy
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- HistoSonics Edison System
  Interventions: Device: HistoSonics Edison System

INTERVENTIONS:
Device: HistoSonics Edison System — Histotripsy with the HistoSonics Edison System for the full or partial destruction of liver tumors
  Other Names: Histotripsy

SUMMARY:
The goal of this observational study is to collect information on the use of the HistoSonics Edison System for the treatment of liver tumors. The main aim is to understand how different patient characteristics and procedural characteristics may affect histotripsy success at 36 hours post-histotripsy procedure. Sub-studies to the BOOMBOX: Master Study will investigate specific populations and/or clinical questions with more stringent enrollment criteria, standardized testing criteria, and/or follow-up schedule. Any participant enrolled in the BOOMBOX: Master Study that also qualifies for a sub-study may enroll in the sub-study in parallel; sub-studies will be described in separate sub-study protocols. The BOOMBOX: Master Study will collect information about participants before, during, and after the histotripsy treatment procedure. All participants will be followed per standard clinical follow-up based on each site's clinical practice for up to 5 years after the initial histotripsy procedure or until completion of their follow-up in a sub-study, whichever is longer.

DETAILED DESCRIPTION:
BOOMBOX: Master Study is an observational, single arm, non-randomized, prospective master study. Following histotripsy treatment of liver tumor(s), subjects will undergo imaging ≤36 hours post-histotripsy treatment procedure to determine histotripsy success. Subjects will then be followed per standard clinical follow-up as determined at each site with regular review of adverse event data for up to 5 years or until completion of their follow-up in a sub-study, whichever is longer.

As an observational study, the master protocol does not direct the use of the HistoSonics Edison System towards any specific clinical intent or any specific disease state. Rather, it will uniformly enroll patients and capture real-world standard-of-care data on the usage of the HistoSonics Edison System as implemented by the treating physician on all subjects treated with histotripsy that meet the study criteria and agree to participate in the study. Sub-studies to the master protocol will investigate specific populations and/or clinical questions with more stringent enrollment criteria, standardized testing criteria, and/or follow-up schedule. Any subject enrolled in the master study who also qualifies for a sub-study may enroll in the sub-study in parallel to the master study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥22 years of age
2. Subject has signed the Ethics Committee (EC), or Institutional Review Board (IRB) approved study Informed Consent Form (ICF) prior to any study related tests/procedures and is willing to comply with study procedures and required follow-up assessments
3. Subject's liver tumor(s) can be partially or completely treated with histotripsy

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant or nursing (lactating) during the study period
2. Subject is enrolled in an interventional HistoSonics-sponsored trial
3. Subject has a concurrent condition that, in the investigator's opinion, could jeopardize the safety of the subject or compliance with the protocol

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are 22 years of age or older with a diagnosis of: primary (e.g., HCC, cholangiocarcinoma, angiosarcoma) or metastatic (from other primary cancers) liver cancer, or benign liver tumors (e.g., adenoma).
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Histotripsy Technical Success | ≤36 hours post-histotripsy treatment procedure
  Histotripsy technical success, defined as completion of histotripsy on the target tumor(s) according to the histotripsy treatment plan, assessed by the treating physician on CT or MR imaging at ≤36 hours post-histotripsy treatment procedure. The histotripsy treatment plan will include identification of the intended complete or partial treatment of the tumor(s). The histotripsy treatment zone must provide target tumor coverage greater than or equal to the degree of treatment intended.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Providence St. Jude, Fullerton, California
  - Mission Hospital, Mission Viejo, California
  - Hoag, Newport Beach, California
  - Providence Saint John's Health Center, Santa Monica, California
  - AdventHealth Altamonte Springs, Altamonte Springs, Florida
  - AdventHealth Celebration, Celebration, Florida
  - Lee Health Cancer Institute, Fort Myers, Florida
  - Baptist Health Miami Cardiac & Vascular Institute, Miami, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - RUSH University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Willis Knighton Health, Shreveport, Louisiana
  - Henry Ford Health, Detroit, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Renown Regional Medical Center, Reno, Nevada
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. David's Medical Center, Austin, Texas
  - Henrico Doctors' Hospital, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No